CLINICAL TRIAL: NCT05543915
Title: Intra-Individual Variability in Cognitive Performance as a Marker of Prodromal Disability in MS
Brief Title: Cognitive Markers in Prodromal MS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Multiple Sclerosis Society (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 21-01385
Record Dates: First submitted 2022-09-13; First posted 2022-09-16 (Actual); Results first posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-06

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Group with tDCS-MRI (Experimental): Participants will have a cognitive assessment, an optional gait assessment, and a 1-hour MRI brain scan combined with 20 minutes of simultaneous tDCS. Participants may also complete the MRI on a separate visit.
  Interventions: Device: Active tDCS
- Group without tDCS- MRI (No Intervention): Participants will have include a cognitive assessment and an optional gait assessment

INTERVENTIONS:
Device: Active tDCS — The tDCS-MRI scan will last approximately one hour. The first 20 minutes of the MRI will not include tDCS stimulation. After 20 minutes, the tDCS device will ramp up to 2.0mA and deliver 2.0mA for 20 minutes. Then the tDCS will ramp down (30 seconds) and the final 20 minutes will be without stimulation.
  Arms: Group with tDCS-MRI

SUMMARY:
The focus of this work is the evaluation of a measure of cognitive functioning- intra-individual variability (IIV) - derived from a computer-based continuous reaction time (RT) task (Cogstate) as an early marker of prodromal MS.

DETAILED DESCRIPTION:
This study is a prospective observational clinical study, where the researchers will recruit adults with early MS (n=60) to complete a cognitive assessment and an optional gait assessment using Runscribe and G-sensor. Thirty-five [35] participants will also have a single 60-minute investigational MRI combined with 20 minutes of simultaneous tDCS. The MRI will repeat the protocol from the researchers' current study (ClinicalTrials.gov Identifier: NCT03564496, IRB i18-00548) using simultaneous transcranial direct current stimulation (tDCS) during the imaging acquisition.

ELIGIBILITY:
Inclusion Criteria:

* Ages 23-59 years old (inclusive)
* Prodromal MS (defined by radiologically isolated syndrome ≤ 6 months from first MRI or clinically isolated syndrome ≤ 3 months from first clinical event)

Exclusion Criteria:

* Below average estimated premorbid cognitive functioning (based on WRAT-4 reading recognition standard z-score < 85).
* Presence of severe cognitive impairment (based on SDMT age normative z-score <-3.0).
* Primary psychiatric disorder that would influence ability to participate.
* Current uncontrolled seizure disorder.
* Current substance abuse disorder.
* History of head trauma in the past year (e.g., head injury, brain surgery) or medical device implanted in the head (such as Deep Brain Stimulator) or in the neck (such as a Vagus Nerve Stimulator).
* Pregnant or breastfeeding

Additional Exclusion Criteria for tDCS-MRI Participants

* Extreme claustrophobia
* Any skin disorder/sensitive skin (e.g., eczema, severe rashes), blisters, open wounds, burn including sunburns, cuts or irritation, or other skin defects which compromise the integrity of the skin at or near stimulation locations (where electrodes are placed)
* Treatment for a communicable skin disorder currently or over the past 12 months
* Have any irremovable piercings, metallic based-tattoos, or MRI-contraindicated implants (e.g. pacemakers and defibrillators)

Ages: 23 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-02-09 (Actual); Primary Completion 2024-06-20 (Actual); Study Completion 2024-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leigh Charvet, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group With tDCS-MRI | Group Without tDCS- MRI
Started | 30 | 30
Completed | 30 | 29
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group With tDCS-MRI | Group Without tDCS- MRI | Total
Number analyzed (Participants) | 30 | 29 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 34 (8.3) | 37 (8.7) | 36 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 23 | 45
  Male | 8 | 6 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 3 | 22
  Not Hispanic or Latino | 5 | 19 | 24
  Unknown or Not Reported | 6 | 7 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 4 | 14
  White | 12 | 16 | 28
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 8 | 9 | 17
Region of Enrollment [Number; unit: participants]
  United States | 30 | 29 | 59

OUTCOME MEASURES:

1. Primary Outcome: Cerebral Metabolic Rate of Oxygen (CMRO2)
Description: CMRO2 is the amount of O2 the brain consumes per unit of time (in μmol O2/100g tissue per minute). To quantify absolute CMRO2, both TRUST MRI for quantification of venous oxygenation (Yv) and phase contrast (PC) MRI for quantification of total blows are needed. The total scan time for CMRO2 MRI is approximately 4 minutes.
Time Frame: Day 1 (Visit 1 - approximately 4 minutes)
Population: Note - assessed in the "Group with tDCS-MRI" arm only.
Measure: Mean (Standard Deviation); unit: micro-mol/100g/min
Arm/Group | Group With tDCS-MRI | Group Without tDCS- MRI
Number analyzed (Participants) | 29 | 0
micro-mol/100g/min | 8.17 (12.99) |

2. Primary Outcome: Intra-Individual Variability (IIV) as Measured by Cogstate Brief Battery (CBB)
Description: The core Cogstate Reaction Time (RT) tasks involve a deck of cards on a green background screen and the participant answers "yes" or "no" by hitting a keyboard key ("D" or "K") across repeated trials. Each task first includes instructions and practice period before the test begins and takes approximately 3-4 minutes to complete (for a total of ~7 minutes). The representative timed RT scores are provided by the Detection task (indicating when a card is revealed; DET/simple RT), Identification task ("is the card revealed black or red?"; IDN/choice RT), and One-Back ("Is this the card that you just saw?"). Performance is characterized by near complete accuracy (i.e. all, or almost all, items are answered correctly), and validity checks are built into the scoring. IIV is calculated as intraindividual standardized deviations (ISD) in RTs across both tasks, measured in milliseconds and with log10 transformation.
Time Frame: Day 1 (Visit 1)
Measure: Mean (Standard Deviation); unit: log10(ms)
Arm/Group | Group With tDCS-MRI | Group Without tDCS- MRI
Number analyzed (Participants) | 30 | 29
log10(ms) | 0.37 (0.64) | 0.34 (0.64)

3. Secondary Outcome: Brief International Cognitive Assessment for MS (BICAMS) Symbol Digit Modalities Test (SDMT) Z-Score
Description: SDMT is 90-second cognitive task in which the participant is shown a sheet containing rows of symbols. Each symbol corresponds to a specific number. The participant's task is to say out loud the number associated with each symbol. SDMT is used as a general cognitive screen to detect severe cognitive impairment. The raw score is the correct number of substitutions in 90 seconds, scores range between 0 and 110. The lower the score, the more severe the cognitive impairment. The raw score is converted to a Z-score with a central value of 0. Standard deviations below the mean indicate a worse outcome; a Z-score of -1.5 or lower suggests a significant deviation from the average performance, potentially indicating cognitive impairment.
Time Frame: Day 1 (Visit 1)
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Group With tDCS-MRI | Group Without tDCS- MRI
Number analyzed (Participants) | 30 | 29
Z-score | -1.09 (1.25) | -1.03 (1.28)

4. Secondary Outcome: BICAMS Rey Auditory Verbal Learning Test (RAVLT) Z-Score
Description: RAVLT is a well-recognized measure of a person's ability to encode, combine, store and recover verbal information in different stages of immediate memory. consists of presenting a list of 15 words across consecutive trials. The list is read aloud to the participant, and then the participant is immediately asked to recall as many words as one remembers. This procedure is repeated for 5 consecutive trials (Trials 1 to 5). The total score is the sum of trials 1-5 and ranges from 0-75. The lower the score, the more severe the cognitive impairment. The raw score is converted to a Z-score with a central value of 0. Standard deviations below the mean indicate a worse outcome; a Z-score of -1.5 or lower indicates impairment, meaning the individual's performance is significantly below the average of their peer group.
Time Frame: Day 1 (Visit 1)
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Group With tDCS-MRI | Group Without tDCS- MRI
Number analyzed (Participants) | 30 | 29
Z-score | -0.17 (0.87) | -0.25 (0.91)

5. Secondary Outcome: BICAMS Brief Visuospatial Memory Test Revised (BVMT-R) Z-Score
Description: Visual/spatial memory is assessed in BICAMS using the BVMT-R. In this test, six abstract designs are presented for 10 sec. The display is removed from view and patients render the stimuli via pencil on paper manual responses. Each design receives from 0 to 2 points representing accuracy and location. There are three Learning Trials, and the score is reported as the total number of points earned over the trials. Thus, scores range from 0 to 12 per trial; total score range is 0 to 36 for all three trials. The lower the score, the more severe the cognitive impairment. The raw score is converted to a Z-score with a central value of 0. Standard deviations below the mean indicate a worse outcome; a Z-score of -1.5 or lower on the BVMT-R is generally considered indicative of cognitive impairment.
Time Frame: Day 1 (Visit 1)
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Group With tDCS-MRI | Group Without tDCS- MRI
Number analyzed (Participants) | 30 | 29
Z-score | 0.14 (1.33) | -0.02 (0.85)

ADVERSE EVENTS:
Time Frame: 1 day (during baseline session).
Description: Participant self-report.
Arm/Group | Group With tDCS-MRI | Group Without tDCS- MRI
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/29
Other Adverse Events (participants affected / at risk) | 1/30 | 0/29
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group With tDCS-MRI (N=30) | Group Without tDCS- MRI (N=29)
Localized warmth sensation at the electrode site (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-04): https://cdn.clinicaltrials.gov/large-docs/15/NCT05543915/Prot_SAP_000.pdf